CLINICAL TRIAL: NCT06522464
Title: Effects Of Modified Constraint Induced Movement Therapy With And Without Cross Education On Upper Limb Function In Cerebral Palsy
Brief Title: Modified Constraint Induced Movement Therapy With And Without Cross Education In Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0772
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Cross education; Modified Constraint-induced; Movement Therapy; dexterity function.
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial in which non probability convenient sampling will be used. Two groups of age 6 - 12 years old CP hemiparetic children having the ability to grasp and release light objects, with an extension of at least 20° of the wrist and 10° of the metacarpophalangeal joints of the fingers (from full flexion of the affected hand will be formed in which participants will be randomly divided. Group A will follow the mCIMT Protocol with additional cross education will be given and group B will follow the mCIMT Protocol.
Who Masked: Investigator
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: mCIMT with cross-education (Experimental): For ten weeks, Group A will follow the mCIMT Protocol, which entails 30 minutes of one-on-one therapy three days a week and five hours a day (weekdays) of constraint.
  In addition, the student will receive extra cross-education, which will involve practicing reaching tasks, wrist flexion and extension, and non-paretic hand opening and closing for 30 minutes. Activities include building a tower out of cubes in various colors, sorting cubes of similar colors and forms together (square cubes in a column, cylindrical cubes together), gripping a hammer, and various cube and triangular shapes. putting balls in their column, placing various-sized circular forms in their proper locations, and moving items between both hands. We'll utilize weight cuffs for every activity.
  Interventions: Other: Group A: mCIMT with cross-education
- Group B: mCIMT without cross-education (Active Comparator): For ten weeks, Group B will follow the mCIMT Protocol, which entails 30 minutes of one-on-one therapy three days a week and five hours a day (weekdays) of confinement.
  Interventions: Other: Group B: mCIMT without cross-education

INTERVENTIONS:
Other: Group A: mCIMT with cross-education — For ten weeks, Group A will follow the mCIMT Protocol, which entails 30 minutes of one-on-one therapy three days a week and five hours a day (weekdays) of constraint.
  In addition, the student will receive extra cross-education, which will involve practicing reaching tasks, wrist flexion and extension, and non-paretic hand opening and closing for 30 minutes. Activities include building a tower out of cubes in various colors, sorting cubes of similar colors and forms together (square cubes in a column, cylindrical cubes together), gripping a hammer, and various cube and triangular shapes. putting balls in their column, placing various-sized circular forms in their proper locations, and moving items between both hands (18). We'll utilize weight cuffs for every activity.
  Arms: Group A: mCIMT with cross-education
Other: Group B: mCIMT without cross-education — For ten weeks, Group B will follow the mCIMT Protocol, which entails 30 minutes of one-on-one therapy three days a week and five hours a day (weekdays) of confinement.
  Arms: Group B: mCIMT without cross-education

SUMMARY:
A nonprogressive injury to the growing brain, cerebral palsy can impair a child's speech, intellectual ability, and motor development. The kind of impairment will correspond with the affected brain region. Cross education is the process of improving one's strength or skill on the contralateral limb after undergoing unilateral training or practice. This is typically done with a mirror, which activates the mirror neuron on the ipsilateral side. CI, or Constraint-Induced Movement Therapy (CIMT), is a "rehabilitative strategy". It is intended to help people affected by stroke or other neurological problems utilize an affected extremity more functionally. It restrains the limb that is neurologically stronger while applying mass practice concepts. It has also been described as a behavioral approach to neurorehabilitation, with a focus on shaping as a recurring theme, and it uses basic behavioral approaches. The study's objective is to ascertain how cross-education using mCIMT affects cerebral palsy that is hemiparetic.

The Pakistan Society for the Rehabilitation of the Disabled, Lahore (PSRD), Rising Sun Institute for Special Children DHA, and ARK campus Lahore will all provide data for the present study, which is a randomized controlled experiment. Twenty-two volunteers will be randomly assigned to two equal groups for the study. Children with hemiperatic cerebral palsy, aged 6 to 12, of any gender, who have up to 20 degrees of wrist extension, 10 degrees of thumb abduction, and up to 10 degrees of finger extension are eligible to participate in the study. Exclusion criteria included significant shoulder subluxation, uncontrolled systemic hypertension, prior stroke, severe heart failure, and a mini mental state evaluation score of less than 24. The control group will receive conventional physical therapy, whereas the experimental group will receive cross-training using mCIMT and RPT. Result The results before and after the intervention will be analyzed using the Fugl Meyer Upper Extremity Scale and Upper Extremity Functional Index Scale, Jebsen-Taylor Hand Function Test, and Block and Box manual Dexterity Test. Data analysis will be conducted using SPSS version 23.00.

DETAILED DESCRIPTION:
Group A:

For ten weeks, Group A will follow the mCIMT Protocol, which entails 30 minutes of one-on-one therapy three days a week and five hours a day (weekdays) of constraint.

In addition, the student will receive extra cross-education, which will involve practicing reaching tasks, wrist flexion and extension, and non-paretic hand opening and closing for 30 minutes. Activities include building a tower out of cubes in various colors, sorting cubes of similar colors and forms together (square cubes in a column, cylindrical cubes together), gripping a hammer, and various cube and triangular shapes. putting balls in their column, placing various-sized circular forms in their proper locations, and moving items between both hands (18). We'll utilize weight cuffs for every activity.

Group B:

For ten weeks, Group B will follow the mCIMT Protocol, which entails 30 minutes of one-on-one therapy three days a week and five hours a day (weekdays) of confinement.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - 12 years old CP hemiparetic children
* having the ability to grasp and release light objects, with an extension of at least 20° of the wrist and 10° of the metacarpophalangeal joints of the fingers (from full flexion of the affected hand)
* having impairment of hand function at levels I to III of the Manual Activity Classification System (MACS)(14).

Exclusion Criteria:

* having visual or auditory disorder
* being subject to seizures or having health problems not associated with CP
* having predominant spasticity or contracture grades more than Grade 3 of the Modified Ashworth Scale in wrist and finger flexors, forearm pronators, and/or thumb adductors
* having received Botulinum neurotoxin injections and/or surgical interventions in the 6-month period before the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Functional Index Scale: | 10 weeks
  Patients with disabilities to their upper limbs can have their functional limitations evaluated using the UEFI. It can be used to track changes in functional status over time and assess how well treatment plans are working. Currently, UEFI 20-item and UEFI 15-item are the two versions available. The UEFI is designed to be used by people who have musculoskeletal dysfunction of the upper extremities (shoulder, elbow, wrist, and hand). The scores on the UEFI range from 0 to 4, where 0 denotes extreme difficulty and 4 denotes no difficulty at all. The total score is the sum of the individual scores. The possible range for the UEFI 20-item is 0 to 80, where 80 represents the highest functioning state and 0 the lowest.
Jebsen-Taylor Hand Function Test: | 10 weeks
  This standardized and objective test uses simulated activities of daily living (ADL) to assess fine and gross motor function in the hands. Writing, simulated page flipping, lifting tiny things, simulated feeding, stacking, and lifting large, light, and heavy objects are the seven subsets of the JTHFT. It is an accurate instrument for measuring hand dysfunctions in a range of patient demographics. The JTHFT takes 15 to 45 minutes to complete. Better performance is shown by shorter times.
Box and Block Test (BBT): | 10 weeks
  The BBT is made up of 150 blocks and a wooden box with a partition dividing it into two sections. requesting that the client transfer the greatest number of blocks, one by one, in 60 seconds from one box compartment to another of equal size. It is especially appropriate for kids for a number of reasons. First, the BBT assessment approach looks at basic manual dexterity skills for growing kids, like gripping, holding, transferring, and releasing. Second, the BBT's instructions are straightforward to understand, and the task itself is simple. Third, the job may be completed in just one minute, which is appropriate for the majority of children's attention spans.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, BS-PT, Principal Investigator — Riphah International University Lahore
Locations (1):
- Rich Care A Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones MW, Morgan E, Shelton JE, Thorogood C. Cerebral palsy: introduction and diagnosis (part I). J Pediatr Health Care. 2007 May-Jun;21(3):146-52. doi: 10.1016/j.pedhc.2006.06.007. PMID 17478303
- [Background] Zulu O, Lupenga J, Simpamba MM, Banda MC. Efficacy of Constraint Induced Movement Therapy and Mirror Therapy in Improving Upper Extremity Function in Late Subacute and Chronic Stroke Patients: A randomized crossover trial. Journal of Preventive and Rehabilitative Medicine. 2023;5(2):136-45.
- [Background] Green LA, Gabriel DA. The cross education of strength and skill following unilateral strength training in the upper and lower limbs. J Neurophysiol. 2018 Aug 1;120(2):468-479. doi: 10.1152/jn.00116.2018. Epub 2018 Apr 18. PMID 29668382